CLINICAL TRIAL: NCT04193475
Title: Machine Learning in Quantitative Stress Echocardiography
Acronym: MLQSE
Status: Recruiting | Type: Observational
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: Barts & The London NHS Trust (Other); Cardiff and Vale University Health Board (Other Government)
Responsible Party: Sponsor
Other Study IDs: R2458
Record Dates: First submitted 2019-11-18; First posted 2019-12-10 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Diseases; Ischaemic Heart Disease
Keywords: Chest pain; Angina; Deformation imaging; Tissue doppler imaging; Strain; Velocity
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Chest Pain; Angina Pectoris; Sprains and Strains

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chest pain: Individuals presenting with chest pain requiring a stress echocardiogram.
  Interventions: Other: Analysis

INTERVENTIONS:
Other: Analysis — No intervention planned. Novel analysis of echocardiographic data.

SUMMARY:
Greater diagnostic accuracy is required to find out who is at risk of a heart attack as this can reduce the requirement of more invasive downstream tests and thereby improve the patient experience and also reduce their exposure to risk. Stress echocardiography is a routine clinical test that involves using ultrasound to image the heart whilst it is under stress to assess the risk of a heart attack.

This study will focus on developing more accurate analysis tools to interpret the results of these stress echocardiographic scans. New methods will be tested to measure the function of each part of the heart muscle, using advanced analysis of the information obtained when high-frequency sound waves are bounced off the heart inside the chest. The researchers will measure and report exact heart function during stress, so that they will be able to recognise normal hearts and those with any disease. New computer methods will be developed to display any abnormality, which will make it easier for doctors to choose the best treatment for patients who are at risk.

The goals and potential benefits of this research proposal are to update the interpretation of a routinely used clinical test (stress echocardiography) to produce a reliable new method for diagnosing the precise effects of diseased arteries on the function of the heart muscle; to develop new computer graphics that adapt to show individual risks for each patient; and to implement new computer models that can be constantly updated

DETAILED DESCRIPTION:
New onset chest pain is a common presenting complaint and can be a marker of significant cardiovascular disease and risk of myocardial infarction and death; therefore obtaining an accurate diagnosis is critical to guide patient management. It is noteworthy that only 40-50% of patients who have invasive arteriography subsequently undergo revascularisation. This underscores the imprecision of the initial tests employed prior to arteriography.

Historically electrocardiographic stress testing during exercise has been used to detect inducible myocardial ischaemia but its diagnostic sensitivity and specificity are low (about 65%). Diagnostic accuracy can be improved by by incorporating echocardiography or single photon emission computed tomography. Current NICE guidelines recommend that patients with chest pain of recent onset should be investigated with CT coronary angiography as a first line, and if this reveals a significant stenosis then a functional imaging test should be performed.

The Myocardial Doppler in Stress Echocardiography (MYDISE) study assessed the diagnostic value of quantitative stress echocardiography during the infusion of dobutamine, a short-acting synthetic catecholamine that acts on β-1 adrenergic receptors to increase heart rate and myocardial contractility. Measuring the systolic velocities of LV long-axis function at peak stress had good reproducibility (coefficients of variation in basal segments 9-14% at rest and 11-18% at peak stress) and similar sensitivities and specificities (about 70%) to published studies in which expert observers reported wall motion scores. When adjusted for the independent effects of age, gender and heart rate, however, diagnostic accuracy increased significantly with C statistics (area under receiver-operator curves) up to 90%.

Visual analysis of stress echocardiography to detect myocardial ischaemia depends on qualitative assessment of multiple parameters. Major studies of quantitative stress echocardiography have been limited to identifying the single best echocardiographic variable, and they have used diameter stenosis as the reference criterion. Progressive subclinical reductions of regional (long-axis) myocardial function have been demonstrated in subjects with cardiovascular risk factors, affecting myocardial deformation (strain and strain rate) as well as velocities. Ischaemia changes the timing of events during the cardiac cycle - for example prolonging pre-ejection and post-ejection phases. These factors confirm the clinical need for objective measurement of regional myocardial function throughout the cardiac cycle.

It is now possible to create algorithms that are based not just on a single time point (e.g., peak velocity) but instead rely on analysis of the whole of the velocity trace. This concept can also be extended to include strain and strain rate curves. Investigators at Universitat Pompeu Fabra, Barcelona, have developed this approach to create a statistical atlas of the heart to detect dyssynchrony. A similar concept has been applied using multiple kernel learning to patients with dyspnoea who have undergone exercise stress testing to identify those with evidence of diastolic heart failure.This has enabled velocity traces taken from the whole of the cardiac cycle to be compared and discriminated between control subjects (with and without dyspnoea) and those diagnosed with heart failure with preserved ejection fraction (HFpEF); the major differences observed are in early diastolic function. This application has not previously been used to explore inducible myocardial ischaemia in stress echocardiography, but similar findings might be expected, as changes during diastole are amongst the earliest and most sensitive indicators of myocardial ischaemia. Individuals at the University of Leuven (Prof Jan D'hooge) have recently developed supervised machine-learning methods that allow for automatic classification of myocardial segments based on their local mechanical behaviour (i.e. velocity/strain/strain rate) after going through a training phase; the proposed machine-learning approach outperforms expert wall motion readings as well as expert interpretation of segmental strain (rate) traces in classifying ischemic segments.

ELIGIBILITY:
Inclusion Criteria:

* Clinically suitable for stress echocardiography examination

Exclusion Criteria:

* None

Ages: 20 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients will be recruited into this study as a single group, with an age range of 20 - 89 years and with no restriction according to their pre-test probabilities of coronary artery disease. They will be eligible for inclusion so long as they have chest pain or another clinical indication for stress testing.
Sampling Method: Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2019-11-22 (Actual); Primary Completion 2025-08-13 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Inducible myocardial ischaemia | 3 years
  Diagnostic performance of the machine learning classifier for the detection of inducible myocardial ischaemia as determined by reduced coronary flow reserve

SECONDARY OUTCOMES:
Workload | 3 years
  Diagnostic performance of workload (units = watts) for the detection of inducible myocardial ischaemia as determined by reduced coronary flow reserve.
Velocity | 3 years
  Diagnostic performance of velocity (units = m/s) for the detection of myocardial functional reserve compared with quantitative coronary arteriography and with coronary flow reserve.
Strain rate | 3 years
  Diagnostic performance of strain rate (units = s^-1) for the detection of myocardial functional reserve compared with quantitative coronary arteriography and with coronary flow reserve.
Strain | 3 years
  Diagnostic performance of strain (units = s) for the detection of myocardial functional reserve compared with quantitative coronary arteriography and with coronary flow reserve.

CONTACTS AND LOCATIONS:
Locations (1):
- Castle Hill Hospital, Cottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided